CLINICAL TRIAL: NCT06671704
Title: GC-PRO Intervention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: CBS-2024-33212
Record Dates: First submitted 2024-10-21; First posted 2024-11-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Cardiovascular Diseases; Prenatal Condition; Reproductive Condition; Genetic Condition
Keywords: genetic counseling; cancer; heart disease; reproductive; prenatal; genetic
MeSH Terms: conditions — Neoplasms; Cardiovascular Diseases; Genetic Diseases, Inborn; Heart Diseases

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cluster 1 (Experimental): Patients recruited and randomized to transfer from standard of care to genetic counselling in months 4-15
  Interventions: Other: Genetic counseling months 4-15
- Cluster 2 (Experimental): Patients recruited and randomized to transfer from standard of care to genetic counselling in months 6-15
  Interventions: Other: Genetic counseling months 6-15
- Cluster 3 (Experimental): Patients recruited and randomized to transfer from standard of care to genetic counselling in months 8-15
  Interventions: Other: Genetic counseling months 8-15
- Cluster 4 (Experimental): Patients recruited and randomized to transfer from standard of care to genetic counselling in months 10-15
  Interventions: Other: Genetic counseling at months 10-15
- Cluster 5 (Experimental): Patients recruited and randomized to transfer from standard of care to genetic counselling in months 12-15
  Interventions: Other: Genetic counseling at months 12-15
- Cluster 6 (Experimental): Patients recruited and randomized to transfer from standard of care to genetic counselling in months 14-15
  Interventions: Other: Genetic counseling at months 14-15

INTERVENTIONS:
Other: Genetic counseling months 4-15 — all genetic counselors within the same specialty at the same site will cross over from standard of care to the intervention training starting at month 4 to month 15.
  Arms: Cluster 1
Other: Genetic counseling months 6-15 — all genetic counselors within the same specialty at the same site will cross over from standard of care to the intervention training starting at month 6 to month 15.
  Arms: Cluster 2
Other: Genetic counseling months 8-15 — all genetic counselors within the same specialty at the same site will cross over from standard of care to the intervention training starting at month 8 to month 15.
  Arms: Cluster 3
Other: Genetic counseling at months 10-15 — all genetic counselors within the same specialty at the same site will cross over from standard of care to the intervention training starting at month 10 to month 15.
  Arms: Cluster 4
Other: Genetic counseling at months 12-15 — all genetic counselors within the same specialty at the same site will cross over from standard of care to the intervention training starting at month 12 to month 15.
  Arms: Cluster 5
Other: Genetic counseling at months 14-15 — all genetic counselors within the same specialty at the same site will cross over from standard of care to the intervention training starting at month 14 to month 15.
  Arms: Cluster 6

SUMMARY:
The goal of the GC-PRO study is to try to make genetic counseling better for people of all backgrounds. We are asking participants to complete two surveys and to allow audio recording of their genetic counseling visit. The purpose of the study is to understand whether trying different ways of doing genetic counseling will lead to better experiences for patients. The research team is also working with partners from the Somali, Latino/Hispanic, Black/African American, and Hmong communities to make sure the research is being done in a way that will benefit underserved communities.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* individual OR their child has been referred to genetic counseling for family and/or personal history of hereditary cancer, cardiology condition, general genetics indication, or reproductive/prenatal indication at a participating study site
* understand and be able to provide information for study forms and surveys in English.

Exclusion Criteria:

* Unable to provide informed consent
* For pediatric genetic counseling referrals, individuals who are not the parent or legal guardian of the child will be excluded from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 994 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
effectiveness of a genetic counseling skills training intervention | 1 month
  The exact measure of effectiveness has been omitted to ensure no bias is created and that research integrity is preserved

SECONDARY OUTCOMES:
patient perception of overall GC quality | 1 month
  Overall perception of quality of the genetic counseling session
patient-centered communication | 1 month
  An assessment of the patient's experience with their healthcare provider
patient empowerment | 1 month
  A process through which patients gain control over decisions and actions affecting their health
patient activation | 1 month
  A patient's ability to manage their own health and take an active role in their care
patient information needs met / information overload | 1 month
  Assessment of how much information the patient desired and was provided
patients' perceived trust in GC | 1 month
  Measure of patients' trust in their provider
working alliance | 1 month
  Relationship between patient and provider
GC verbal dominance | 1 month
  Measurement of the amount of time the patient, genetic counselor, and other individuals spend talking in the session

CONTACTS AND LOCATIONS:
Overall Officials: Heather Zierhut, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States